CLINICAL TRIAL: NCT05416034
Title: Study of the Impact of a Gait Exoskeleton on the Quality of Life of Patients With Spinal Muscular Atrophy
Brief Title: Exoskeleton Impact on the Quality of Life on Patients With Spinal Muscular Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KINDER
Record Dates: First submitted 2022-05-03; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Spinal Muscular Atrophy Type II
Keywords: exoskeleton; spinal muscular atrophy; care; quality of life; robotics
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of the ATLAS 2030 exoskeleton at home (Experimental): Children with Spinal Muscular Atrophy Type II will received robot assisted gait therapy with the ATLAS 2030 exoskeleton at their homes 5 days a week during two months in 60 minutes sessions
  Interventions: Device: Use of the ATLAS 2025 exoskeleton at home

INTERVENTIONS:
Device: Use of the ATLAS 2025 exoskeleton at home — Each participant will use the ATLAS 2025 exoskeleton at their homes, 5 days a week during a period of two months, for walking with the device and performing motor activities in 60 minutes duration sessions..

SUMMARY:
The purpose of this study is to evaluate the impact of the use of a pediatric exoskeleton on the quality of life of children, specifically in the psychological and care dimensions. Other objectives are to evaluate changes at the physical and functional level.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 4 and 9 years old
* Patients with a confirmed diagnostic of Spinal Muscular Atrophy Type II

Exclusion Criteria:

* Weight over 40 Kg
* Hip-knee distance less than 22 cm or greater than 38cm
* Knee-ankle distance less than 21 cm or greater than 37cm
* Distance between trochanters less than 24 cm or greater than 40cm
* Joint range limit greater than 20º

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Phenomenological Interviews | 2 months
  Assess the psychological impact of the experience on both children and the main care giver through phenomenological interviews.
  The phenomenological interview was an open interview evaluating how the participants lived the experience of using an exoskeleton at home
Care impact | 2 months
  To evaluate the impact of the experience in self-care of children by conducting nursing evaluations based on the Self-Care Theory developed by Dorothea Orem, before, during the use of the exoskeleton and at the end. To collect the data needed to complete the nursing assessment, structured nursing interviews were conducted with each child's primary caregiver.
  No scales are used to assess the care impact. A positive care impact will be considered if by using the exoskeleton any children or parents have an increase in any self-care agency.
  A negative care impact will be considered if by using the exoskeleton any self-care demand can not be satisfied by the self-care agency of any of the children or parents.
Participant observation | 2 months
  Assess the psychological impact of the experience on both children and the main care giver through participant observation.
  Participant observation was performed during exoskeleton use sessions in the children's homes. Data was taken by field notes of everything that happened during the session.

SECONDARY OUTCOMES:
Upper limb Function | 2 months
  Assessed by the Revised Upper Limb scale used to investigate the upper limb function of ambulatory and nonambulatory patients with Spinal Muscular Atrophy. The scale has 19 scorable items// Each item is scored from 0 to 2 0=Unable 1=Able, with modiﬁcation 2=Able, no difﬁculty. The best possible final score is 0 and the worst final possible score is 38.
Number of Steps | 2 months
  Changes in the physical performance with the exoskeleton of the children over time by assessing the number of steps. This data collected directly from the device information.
Muscle Strength | 2 months
  Changes in muscle strength over time assessed by a hand held dynamometer at the begginig and at the end of the study. Every lower limb muscle is measured 3 times and the best result of the 3 is taken.
Number of participants with abnormal vital signs | 2 months
  The data obtained in vital signs before and after using the exoskeleton will be analysed by comparing the data with the Pediatric Emergency Assessment Recognition and Stabilization (PEARS) Vital Signs form the American Heart Association. Any abnormal value will be registered.
Respiratory rate (breaths/min) | 2 months
  The therapist took the respiratory rate by counting the number of breaths in one minute by observing the movement of the chest as the child breathed, before and after each session.
Oxygen saturation | 2 months
  Oxygen saturation and heart rate were measured with a suitable pediatric pulse oximeter using the PC-900PRO® (Creative Medical®, Shenzen, China) before and after each session.
Self percieved fatigue | 2 months
  Changes in self percieved fatigue before and after each session by using the OMNI (Omnibus) scale, a developmentally indexed category format that con- tains both pictorial and verbal descriptors positioned along a comparatively narrow numerical response range, i.e. category range 0 to 10. The best possible result is 0 and the worst is 10.
Motor Function | 2 months
  Assessed by the Hammersmith Functional Motor Scale for Spinal Muscular Atrophy. Designed with a 3 point scoring system: Score 2 = performs without modification/adaptation/compensation Score 1 = performs with modification/adaptation/compensation Score 0 = unable to perform Specific scoring criteria per item is outlined in detail in this manual. The best possible final score is 0 and the worst final possible score is 99.
Duration of time walking in each session. | 2 month
  Changes in the physical performance with the exoskeleton of the children over time by recording the duration of time walking in each session. This data collected directly from the device information.
Blood pressure | 2 months
  Systolic and Diastolic blood pressure (mmHg). Using the PC-900PRO® (Creative Medical®, China) before and after each session.
  Blood pressure is taken with the child sitting, always using the same arm for each child, with the correct cuff size and with the arm at heart level.
Social behaviour | 2 months
  Assessed by a semi-structured interview done to the child and the main care giver, and by participant observation which questions are focused on social behaviour aspects.
  No scales were used to assess the sense of agency.
Exploration | 2 months
  Assessed by a semi-structured interview done to the child and the main care giver, and by particpant observation which questions are focused on exploration aspects. .
  Participant observation was performed during exoskeleton use sessions in the children's homes. Data was taken by field notes of everything that happened during the session and the analysis focused on exploration aspects.
  No scales were used to assess exploration.
Sense of agency | 2 months
  Assessed by a semi-structured interview done to the child and the main care giver, and by participant observation which questions are focused on the sense of agency aspects.
  Participant observation was performed during exoskeleton use sessions in the children's homes. Data was taken by field notes of everything that happened during the session and the analysis focused on the sense of agency aspects.
  No scales were used to assess the sense of agency.
Emotional impact | 2 months
  Assessed by a semi-structured interview done to the child and the main care giver which questions are focused on the emotional aspects, and by participant observation.
  Participant observation was performed during exoskeleton use sessions in the children's homes. Data was taken by field notes of everything that happened during the session and the analysis focused on emotional impact aspects.
  No scales were used to assess the emotional impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No